CLINICAL TRIAL: NCT00002520
Title: Brief Physician-Initiated Quit Smoking Strategies for Clinical Oncology Settings
Brief Title: Physician-Initiated Stop-Smoking Program for Patients Receiving Treatment for Early-Stage Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CDR0000078281; U10CA021115 (NIH); E-1Y92; NCI-P93-0042
Record Dates: First submitted 1999-11-01; First posted 2003-08-11 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Bladder Cancer; Breast Cancer; Colorectal Cancer; Head and Neck Cancer; Lung Cancer; Lymphoma; Prostate Cancer; Testicular Germ Cell Tumor; Tobacco Use Disorder; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage I adult Hodgkin lymphoma; angioimmunoblastic T-cell lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage I colon cancer; stage II colon cancer; stage I breast cancer; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; anaplastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; intraocular lymphoma; limited stage small cell lung cancer; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; primary central nervous system lymphoma; tobacco use disorder; stage I adenoid cystic carcinoma of the oral cavity; stage I adult T-cell leukemia/lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult Burkitt lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I basal cell carcinoma of the lip; stage I cutaneous T-cell non-Hodgkin lymphoma; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I lymphoepithelioma of the nasopharynx; stage I lymphoepithelioma of the oropharynx; stage I mantle cell lymphoma; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I mycosis fungoides/Sezary syndrome; stage I non-small cell lung cancer; stage I prostate cancer; stage I rectal cancer; stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I malignant testicular germ cell tumor; stage I verrucous carcinoma of the larynx; stage I verrucous carcinoma of the oral cavity; stage II adult T-cell leukemia/lymphoma; stage II adenoid cystic carcinoma of the oral cavity; stage II basal cell carcinoma of the lip; stage II bladder cancer; stage II breast cancer; stage II cutaneous T-cell non-Hodgkin lymphoma; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II lymphoepithelioma of the nasopharynx; stage II lymphoepithelioma of the oropharynx; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II mycosis fungoides/Sezary syndrome; stage I bladder cancer; stage II non-small cell lung cancer; stage II prostate cancer; stage II rectal cancer; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II malignant testicular germ cell tumor; stage II verrucous carcinoma of the larynx; stage II verrucous carcinoma of the oral cavity; stage III adult T-cell leukemia/lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Burkitt lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage III prostate cancer; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IV adult T-cell leukemia/lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; stage IV prostate cancer; unspecified adult solid tumor, protocol specific; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Lymphoma; Prostatic Neoplasms; Testicular Germ Cell Tumor; Tobacco Use Disorder; Hodgkin Disease; Immunoblastic Lymphadenopathy; Colonic Neoplasms; Lymphoma, Large-Cell, Anaplastic; Intraocular Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Esthesioneuroblastoma, Olfactory; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Carcinoma, Non-Small-Cell Lung; Rectal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Testicular Neoplasms; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quit Smoking Intervention (Experimental): Patients received advice and help to quit smoking. The intervention employed physician and patient resources that had already been developed and evaluated or pre-tested, including written materials, prescriptions for nicotine replacement, counseling, and follow-up contact.
  Interventions: Drug: nicotine
- Usual Care (Active Comparator): No special intervention after randomization. "Usual care" may or may not include advice or assistance to stop smoking. Physicians were reassured that "usual care" did not preclude quit smoking counseling.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Drug: nicotine
  Arms: Quit Smoking Intervention
Behavioral: Usual Care
  Arms: Usual Care

SUMMARY:
RATIONALE: Physician-initiated smoking cessation strategies may be effective in getting early-stage cancer patients to quit smoking.

PURPOSE: Randomized clinical trial to compare the effectiveness of a physician-initiated stop-smoking program with the usual care for patients receiving treatment for early-stage cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of brief physician-initiated smoking cessation strategies vs usual care in patients with early stage cancer who are undergoing treatment in clinical oncology settings.
* Compare the sociodemographic, smoking history, and health status correlates of smoking cessation in patients treated with these regimens.
* Determine the feasibility of conducting a cancer prevention and control study in a cooperative group setting by monitoring adherence to the smoking-cessation strategies.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive usual care (no special intervention).
* Arm II: Patients receive smoking-cessation therapy based on the 4-step intervention plan in the "Manual for Physicians" published by the National Cancer Institute. The smoking cessation coordinator and physician provide self-quitting advice and support to the patient via counseling, self-help materials, and referral to a smoking cessation counselor at the Cancer Information Service (CIS). Patients receive nicotine replacement, if indicated. Patients who express an interest in more intensive treatment are referred to local American Cancer Society or American Lung Association clinics and/or advised to call the CIS for additional local program referrals.

All patients are followed at 6 and 12 months. Patients who report that they are still smoking and interested in help to quit smoking at the 12-month follow-up interview are encouraged to return to their physicians and contact the CIS for additional help quitting or for a referral to more intensive or specialized treatments in their area.

PROJECTED ACCRUAL: A total of 494 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Stage I or II bladder, colorectal, head and neck, lung, or other cancer
  * Stage I-III testicular cancer
  * Stage I-IV breast cancer, prostate cancer, or lymphoma
* Must have smoked 1 or more cigarettes within the past month or define self as a smoker
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 19 and over

Sex:

* Not specified

Menopausal status:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No history of recent heart attack

Other:

* Not pregnant
* No other imminent medical needs requiring referral to a more intensive smoking cessation regimen

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior participation in the pilot phase study

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 1990-12-07 (Actual); Primary Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Rate of Smoking Cessation at 6 months | Assessed at 6 months
  Proportion of patients who have quit smoking 6 months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Paul F. Engstrom, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Schnoll RA, Zhang B, Rue M, Krook JE, Spears WT, Marcus AC, Engstrom PF. Brief physician-initiated quit-smoking strategies for clinical oncology settings: a trial coordinated by the Eastern Cooperative Oncology Group. J Clin Oncol. 2003 Jan 15;21(2):355-65. doi: 10.1200/JCO.2003.04.122. PMID 12525530